CLINICAL TRIAL: NCT04135963
Title: Clinical and Sociodemographic Characterization of Multiple Myeloma Patients With Symptomatic Relapse and/or Refractory Disease in Portugal: an Observational, Multicenter Study
Brief Title: A Study of People With Multiple Myeloma (MM) in Portugal (CharisMMa-Portugal)
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: RRMM-5017; U1111-1234-4861 (Registry Identifier: WHO)
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Relapse and/or Refractory Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with MM: Participants diagnosed with MM from 8 investigative sites will be observed retrospectively for previous 5 years before enrollment until Day 1.

SUMMARY:
The main aim of this study is to see how people with MM respond to previous or current treatment.

Participants will be treated according to their clinic's standard practice. Each participant will fill out a study questionnaire during a routine doctor visit. Information collected from past medical records will also be used.

DETAILED DESCRIPTION:
This is a non- interventional, retrospective epidemiological study of participants with MM. The study will characterize MM participants with symptomatic relapse and/or refractory (R/R) disease.

The study will enroll approximately 151 participants. The study will have a retrospective data collection referring to previous 5 years from participants' records and medical charts regarding diagnosis, disease activity, treatment patterns, and healthcare resources while quality of life (QoL) will be obtained from European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ)-C30 and EORTC QLQ-MY20 questionnaires. All participants will be enrolled in one observational group.

This multi-center trial will be conducted in Portugal. The overall time to participate in this study is limited to completion of a questionnaire at the time of joining the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least one previous treatment line.
2. Symptomatic R/R disease in the previous 6 months to study enrolment.
3. Receiving treatment with an accurate and thorough data fulfilled in their participant's medical records available at the study site.
4. On regular follow-up for relapse and/or refractory disease during the recruitment period at the study site.
5. Capable of understanding and completing both QoL questionnaires (EORTC QLQ-C30 and EORTC QLQ-MY20).

Exclusion Criteria:

1. Diagnosed with MM more than 5 years previous to inclusion in this study.
2. Diagnosed with any malignancy other than MM or its complications within the past 5 years.
3. Currently participating in a clinical trial for his MM or having participated in a clinical trial within 5 years before inclusion.
4. Diagnosed with any hematological disease other than MM or its complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of MM with symptomatic R/R disease receiving treatment in Portugal.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Number of MM Participants Categorized by Sociodemographic Variables | Day 1
  The sociodemographic variables will include age (in years), sex (male or female), body mass index (BMI), area of residence (rural or urban), educational level (illiterate, no studies (can only read/write), primary studies, secondary studies, or university studies), cohabitation (lives alone, lives with the family, lives alone with help from a caregiver, daily, 2-3 times/week, permanent or night-time), degree of dependence (independent, dependent grade I- requires help to perform instrumental activities of daily living (IADL) at least once a day, dependent grade II- needs help to perform IADLs 2 or 3 times a day or dependent grade III- needs help to perform IADLs several times a day),working situation (unemployed, in active employment, temporarily/permanently disabled, retired, student, other, need for financial assistance (yes/no), physical activity (high, moderate/low, inactive), smoking habit (yes/no), alcohol use (yes/no).
Number of MM Participants Categorized by Clinical Variables on Diagnosis and During Previous Relapses | Day 1
  Clinical variables will include age (at diagnosis); MM type; international staging system (ISS) disease stage; Revised-ISS (R-ISS) disease stage; SliMCRAB signs at time of diagnosis: plasma cell bone marrow infiltration greater than or equal to (>=) 60 percent (%), serum free light chain (FLC) ratio >=100, >1 focal lesion visible on magnetic resonance imaging (MRI) with 5 millimeter (mm) or greater, increased blood calcium, renal failure, anemia, bone lesions: one or more osteolytic lesion on standard radiograph, computed tomography (CT) or Positron emission tomography-CT (PET-CT); cytogenetic abnormalities at time of diagnosis (t[4;14], t[11;14], t[14;16], t[14;20], t[6;14], trisomies, d[17p], g[1q]/ others); risk according to cytogenetic profile at diagnosis (mSMART v2 and mSMART v3); previous relapses (before the latest); stem cell transplant (yes/no); eastern cooperative oncology group (ECOG: 0-4) on diagnosis.
Number of MM Participants Categorized by Clinical Variables at Last R/R Episode | Day 1
  Clinical variables include date of latest symptomatic relapse and/or refractory episode; ISS disease stage, CRAB signs; other clinical variables (plasmacytomas: medullary or extramedullary, diffuse osteopenia, fractures, neurological symptoms, infections, lactate dehydrogenase levels, paraprotein levels, free light chain levels); concomitant diseases (diabetes, neuropathy, chronic obstructive pulmonary disease, cardiovascular disease, liver failure, psychiatric and/or neurological disorders, any other secondary disorders); cytogenetic abnormalities at diagnosis; risk according to cytogenetic profile at relapse; treatment started after latest symptomatic relapse and/or refractory episode.
Number of Participants Categorized by Current Treatment | Day 1
  Type of treatment will include therapeutic group.

SECONDARY OUTCOMES:
Number of Participants Categorized by Sociodemographic Characteristics at the Latest Symptomatic R/R Episode per Type of Treatment | Day 1
  Sociodemographic variables will include age (in years), sex (male or female), BMI, area of residence (rural or urban), educational level (illiterate, no studies (can only read/write), primary studies, secondary studies, or university studies), cohabitation (lives alone, lives with the family, lives alone with help from a caregiver, daily, 2-3 times/week, permanent or night-time), degree of dependence (independent, dependent grade I - requires help to perform IADL at least once a day, dependent grade II - needs help to perform IADLs 2 or 3 times a day or dependent grade III - needs help to perform IADLs several times a day), need for financial assistance (yes/no), smoking habit (yes/no), alcohol use (yes/no).
Number of MM Participants Categorized by Clinical Variables at Latest Symptomatic R/R Episode per Type of MM | Day 1
  Clinical variables will include- date of latest symptomatic R/R episode; SLiMCRAB signs at latest symptomatic R/R episode: plasma cell bone marrow infiltration >=60 %, serum FLC ratio >=100, >1 focal lesion visible on MRI with 5 mm or greater, increased blood calcium, renal failure, anemia, bone lesions: one or more osteolytic lesion on standard radiograph, CT or PET-CT; other clinical variables at latest symptomatic R/R episode include- plasmacytomas (medullary/extramedullary); diffuse osteopenia; fractures; neurological symptoms (MM related); infections; lactose dehydrogenase (LDH); paraprotein levels (gram per liter [g/L]) (serum and urine) free light chain levels (g/L) (serum and urine).
Number of Participants Categorized by Relevant Variables that are not Currently Collected in Clinical Record and Could Influence in the Disease Management at Relapse | Day 1
  New relevant variables will include factors mentioned by the participant as relevant to the disease management (example, family support, employment status); type of transportation used to receive treatment; mean cost in Euros per month with transportation to receive treatment, mean of hospital visits per month since last treatment was initiated, mean scheduled and non-scheduled participant's visits to the hospital, days of hospitalization, and specialists consulted; consultations, days of hospitalization, medical appointments and specialists consulted by type of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (8):
- Portugal (8):
  - Centro Clinico Academico Hospital de Braga, Braga
  - Centro Hospitalar e Universitario de Coimbra. EPE, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil (IPO), Lisbon
  - Centro Hospitalar Lisboa Norte EPE - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar Universitario do Porto, E.P.E., Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, E.P.E., Porto
  - Centro Hospitalar Universitario de Sao Joao, EPE,, Porto
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, EPE,, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information about this study, click this link. — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a35f?idFilter=%5B%22RRMM-5017%22%5D